CLINICAL TRIAL: NCT05538767
Title: Efficacy and Safety of Emodepside in Adolescents and Adults Infected With Trichuris Trichiura and Hookworm: Randomized Two Stages Phase II Seamless Adaptive Controlled Single-blind Trials
Brief Title: Efficacy and Safety of Emodepside in Adolescents and Adults Infected With Hookworm
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jennifer Keiser (Other)
Collaborators: Public Health Laboratory Ivo de Carneri (Other)
Responsible Party: Sponsor-Investigator, Jennifer Keiser, Prof. Dr., Swiss Tropical & Public Health Institute
Organization: Swiss Tropical & Public Health Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMODEPSIDE_PEMBA
Record Dates: First submitted 2022-09-09; First posted 2022-09-14 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Hookworm Infections
Keywords: Hookworm; Emodepside; Efficacy; Safety; Confirmatory Stage; Soil Transmitted Helminth
MeSH Terms: conditions — Hookworm Infections; Ancylostomiasis | interventions — emodepside; Albendazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emodepside 30 mg (Experimental)
  Interventions: Drug: Emodepside
- Albendazole 400 mg (Active Comparator)
  Interventions: Drug: Albendazole 400mg

INTERVENTIONS:
Drug: Emodepside — Treatment with Emodepside 30 mg
  Arms: Emodepside 30 mg
Drug: Albendazole 400mg — Treatment with Albendazole 400 mg
  Arms: Albendazole 400 mg

SUMMARY:
To compare the efficacy and safety of emodepside to that of albendazole (Zentel®) in participants aged 12-60, inclusive, infected with hookworm.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged between 12 and 60 years;
* Written and signed informed consent;
* Was examined by a study physician before treatment;
* Provided two stool samples at baseline;
* Hookworm EPG > 48 and at least two Kato-Katz thick smears slides with more than one hookworm eggs.

Exclusion Criteria:

* Pregnant or lactating and/or planning to become pregnant within three months after drug treatment;
* Type 1 and/or 2 diabetes;
* Psychiatric disorders;
* History of ophthalmological conditions;
* Presence or history of major systemic or chronic illnesses, as assessed by a medical doctor, during initial clinical assessment;
* Suffers from severe anaemia (Hb < 80 g/l);
* Received anthelminthic treatment within past four weeks;
* Attending other clinical trials during the study;
* Received strong CYP3A4 inducers or inhibitors as well as concomitant treatments that are relevant substrate for CYP3A4 such as clarithromycin, erythromycin and rifampicin;
* Received strong P-gp inhibitors as well as concomitant treatments that are relevant substrates for P-gp such as clotrimazole and ritonavir.
* Participated in stage I trials of this protocol

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 320 (Actual)
Dates: Start 2022-09-16 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
Cure rate (CR) of emodepside against hookworm | In the week between 14 and 21 days post-treatment
  CR will be calculated as the percentage of hookworm egg-positive participants at baseline who become egg-negative after treatment.

SECONDARY OUTCOMES:
Geometric Mean Egg Reduction Rate (ERR) of the emodepside against hookworm. | In the week between 14 and 21 days post-treatment
  Eggs per gram of stool (EPG) will be assessed by adding up the egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of six. The egg reduction rate (ERR) is calculated as follows: ERR = (1-(geometric mean EPG at follow-up/geometric mean EPG at baseline))*100). Note: in contrast to the publication the "outcome measure" entry mask requires the complementary percentage: (geometric mean at follow-up/geometric mean at baseline)*100).
CR of emodepside against Trichuris trichiura and Ascaris lumbricoides | In the week between 14 and 21 days post-treatment
  CR will be calculated as the percentage of Trichuris trichiura and Ascaris lumbricoides egg-positive participants at baseline who become egg-negative after treatment.
ERR of the emodepside against Trichuris trichiura and Ascaris lumbricoides. | In the week between 14 and 21 days post-treatment
  EPG will be assessed by adding up the egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of six. The ERR is calculated as follows: ERR = (1-(geometric mean EPG at follow-up/geometric mean EPG at baseline))*100). Note: in contrast to the publication the "outcome measure" entry mask requires the complementary percentage: (geometric mean at follow-up/geometric mean at baseline)*100).
Infection status and intensity assessed for at baseline and 14-21 days post-treatment by FECPAK-G2. | At baseline and 14-21 days post-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Public Health Laboratory Ivo de Carneri, Chake Chake, Pemba, Tanzania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Taylor L, Ahmada AA, Ali MS, Ali SM, Hattendorf J, Mohammed IS, Keiser J. Efficacy and safety of emodepside compared with albendazole in adolescents and adults with hookworm infection in Pemba Island, Tanzania: a double-blind, superiority, phase 2b, randomised controlled trial. Lancet. 2024 Aug 17;404(10453):683-691. doi: 10.1016/S0140-6736(24)01403-X. PMID 39153818